CLINICAL TRIAL: NCT04670315
Title: Validation of theTelematic Spanish Version of the Fugl-Meyer Assessment of Motor Recovery After Stroke
Brief Title: Validation of the Telematic Version of the Fugl-Meyer Scale
Status: Completed | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Llamas-Ramos, Associate Professor, University of Salamanca
Other Study IDs: NEUROUSAL03/2020
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Stroke; Validation Study; Patient Outcome Assessment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group: Scale validation in stroke patients
  Interventions: Diagnostic Test: Telematic evaluation of motor function

INTERVENTIONS:
Diagnostic Test: Telematic evaluation of motor function — Validation of the Telematic Spanish Version of the Fugl Meyer Assessment Scale

SUMMARY:
Stroke is one of the most prevalent pathologies worldwide and its consequences require long-term treatment. The current situation caused by the Sars-cov-2 virus has collapsed health systems and has delayed these patient's treatment. The proposed alternative is telerehabilitation: a treatment system that has already proved its effectiveness. However, the difficulty to assess the stroke patient's functional status is the great problem. For this reason, a Fugl Meyer Assessment Scale adaptation, one of the most widely used (in research and in clinic), is proposed to be carried out remotely. The objective of our study is to validate this scale in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18-years-old
* Diagnosis of stroke

Exclusion Criteria:

* Another neurological or orthopedic problem different than stroke that will affect functionality and balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years with a diagnosis of stroke
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment of sensorimotor function | baseline
Fugl-Meyer Assessment Upper Extremity (FMA-UE) | Baseline
Fugl-Meyer Assessment Lower Extremity (FMA-LE) | Baseline
Fugl Meyer Assessment of sensorimotor function (Short Form) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided